CLINICAL TRIAL: NCT05440136
Title: A Single-Ascending Dose, Safety, Tolerability, and Pharmacokinetic Study of LY3462817 in Healthy Japanese and Non-Japanese Participants
Brief Title: A Safety Study of LY3462817 in Healthy Japanese and Non-Japanese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 18141; J1A-MC-KDAE (Other: Eli Lilly and Company)
Record Dates: First submitted 2022-06-27; First posted 2022-06-30 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- LY3462817 - SC (Experimental): LY3462817 administered subcutaneously (SC)
  Interventions: Drug: LY3462817 (SC)
- LY3462817 - IV (Experimental): LY3462817 administered intravenously (IV)
  Interventions: Drug: LY3462817 (IV)
- Placebo - SC (Placebo Comparator): Placebo administered SC
  Interventions: Drug: Placebo (SC)
- Placebo - IV (Placebo Comparator): Placebo administered IV
  Interventions: Drug: Placebo (IV)

INTERVENTIONS:
Drug: LY3462817 (SC) — Administered SC.
  Arms: LY3462817 - SC
Drug: Placebo (SC) — Administered SC.
  Arms: Placebo - SC
Drug: LY3462817 (IV) — Administered IV.
  Arms: LY3462817 - IV
Drug: Placebo (IV) — Administered IV.
  Arms: Placebo - IV

SUMMARY:
The main purpose of this study is to evaluate the safety and tolerability of LY3462817 in healthy Japanese and non-Japanese participants. The study will also assess how fast LY3462817 gets into the blood stream and how long it takes the body to remove it. The study is open to healthy participants. The study will last up to approximately 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy as determined by medical evaluation
* Japanese participants must be first generation Japanese and have a body mass index (BMI) of 18.0 to 30.0 kilograms per square meter (kg/m²) (inclusive), and a body weight of 45 and 85 kg (inclusive)
* Non-Japanese participants have a BMI of 18.0 to 32.0 kg/m² (inclusive), and a minimum body weight of 45 kg
* Are males who agree to follow contraception requirements or females not of childbearing potential
* Have blood pressure, pulse rate, electrocardiogram (ECG, heart tracing), blood and urine laboratory test results that are acceptable for the study

Exclusion Criteria:

* Are currently participating in or completed a clinical trial within the last 30 days or any other type of medical research judged to be incompatible with this study
* Have previously participated or withdrawn from this study
* Have cancer or a malignant disease in the past 5 years
* Have or used to have health problems or laboratory test results or ECG readings that, in the opinion of the doctor, could make it unsafe to participate, or could interfere with understanding the results of the study
* Are unwilling to receive study drug administration by injections or through the veins

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2022-06-28 (Actual); Primary Completion 2023-03-08 (Actual); Study Completion 2023-03-08 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline through Week 12
  A summary of TEAEs, SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC) of LY3462817 | Predose on Day 1 through Day 85
  PK: AUC of LY3462817
PK: Maximum Concentration (Cmax) of LY3462817 | Predose on Day 1 through Day 85
  PK: Cmax of LY3462817

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Altasciences Clinical Los Angeles, Inc, Cypress, California, United States

IPD SHARING:
Plan to Share IPD: No